CLINICAL TRIAL: NCT01766037
Title: Pivotal Aspiration Therapy With Adjusted Lifestyle Therapy Study
Acronym: PATHWAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aspire Bariatrics, Inc. (Industry)
Collaborators: Boston Medical Center (Other); Brigham and Women's Hospital (Other); Cornell University (Other); Howard University (Other); Mayo Clinic (Other); Northwestern University (Other); St. Mary's Medical Center (Other); San Diego Veterans Healthcare System (U.S. Federal Agency); University of Pennsylvania (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P12-001V
Record Dates: First submitted 2013-01-07; First posted 2013-01-11 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Obesity
Keywords: obesity; obese; weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspiration Therapy (Experimental): Aspiration Therapy and Lifestyle Therapy
  Interventions: Device: Aspiration Therapy (AspireAssist); Behavioral: Lifestyle Therapy
- Lifestyle Therapy (Active Comparator): Lifestyle Therapy only
  Interventions: Behavioral: Lifestyle Therapy

INTERVENTIONS:
Device: Aspiration Therapy (AspireAssist) — Use of the AspireAssist device in aspiration therapy
  Other Names: AspireAssist Aspiration Therapy System
  Arms: Aspiration Therapy
Behavioral: Lifestyle Therapy — Lifestyle therapy is a behavioral, diet and physical activity education program
  Other Names: Lifestyle Behavioral Therapy

SUMMARY:
This research study is being performed to find out if a new device, AspireAssist Aspiration Therapy System, can help people with obesity to lose weight without causing too many side effects.

DETAILED DESCRIPTION:
The Aspiration process works by "correcting" meal portions after eating by removing some of the food left in your stomach 20 minutes after your meal, which reduces the number of calories absorbed by your body. This is done through a tube placed through the abdomen into the stomach with a small valve attached at the surface of your skin. An aspiration system will attach to that valve after each major meal of the day and allow you to remove a portion of that meal.

During this study you will also be provided with Lifestyle therapy which includes behavioral therapy, diet and physical activity education. This Lifestyle therapy will also be provided to the participants who do not receive the AspireAssist so that the two groups can be compared and the benefit of aspiration for weight loss can be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Measured BMI of 35.0-55.0 kg/m2 at time of screening.
2. 21- 65 years of age (inclusive) at time of screening.
3. Failed attempt for a duration equal to 3-months at weight loss by alternative approaches (e.g. supervised or unsupervised diets, exercise, behavioral modification programs).
4. Stable weight (<3% change in self-reported weight) over the previous 3 months at time of screening).
5. Women of childbearing potential must agree to use at least one form of birth control (prescription hormonal contraceptives, diaphragm, IUD, condoms with or without spermicide, or voluntary abstinence) from time of study enrollment through study exit.
6. Willing and able to provide informed consent in English and comply with the protocol.

Exclusion Criteria:

1. Previous abdominal surgery that significantly increases the medical risks of gastrostomy tube placement
2. Esophageal stricture, pseudo-obstruction, severe gastroparesis or gastric outlet obstruction, inflammatory bowel disease
3. History of refractory gastric ulcers
4. Ulcers, bleeding lesions, or tumors discovered during endoscopic examination.
5. History of radiation therapy to the chest or abdomen
6. Uncontrolled hypertension (blood pressure >160/100).
7. Diabetes treated with insulin or sulfonylurea medications
8. Any change in diabetes medication in previous 3 months
9. Hemoglobin A1C >9.5%
10. History or evidence of serious pulmonary or cardiovascular disease, including acute coronary syndrome, heart failure requiring medications, or NYHA (New York Heart Association) class III or IV heart failure (defined below):

    Class III: patients with marked limitation of activity and who are comfortable only at rest Class IV: patients who should be at complete rest, confined to bed or chair and who have discomfort with any physical activity
11. Coagulation disorders (platelets < 100,000, PT > 2 seconds above control or INR > 1.5)
12. Anemia (Hemoglobin <11.0 g/dL in women and <12.5 g/dL in men)
13. Liver enzymes (ALT and AST) ≥3.0 times the upper limit of normal
14. Thyroid Stimulating Hormone (TSH) >1.5 x upper limit of normal at screening.
15. Osteoporosis (DEXA T-Score ≤ -2.5 standard deviations below normal peak values).
16. History of fragility fractures (fractures resulting from a fall from a standing height or less, or presenting in the absence of obvious trauma)
17. Pregnant or lactating
18. Diagnosed Bulimia or diagnosed Binge Eating Disorder (using DSM IV criteria)
19. Night Eating Syndrome (diagnosed by EDE)
20. Serum potassium < 3.8 mEq/L
21. Chronic abdominal pain that would potentially complicate the management of the device
22. Taking a GLP-1 agonist < 6 months.
23. Taking prescription or over-the-counter medications for weight loss in the last 3 months before screening, or planning to participate in a commercial weight loss program in the next 24 months.
24. Taking medication once or more per week that causes weight gain (e.g. atypical antipsychotics, monoamine oxidase inhibitors, lithium, selected anticonvulsants, tamoxifen, glucocorticoids)
25. Self- reported history of substance abuse in last 3 years.
26. Malignancy in the last 5 years (except for non-melanoma skin cancer).
27. Physical or mental disability, or psychological illness that could interfere with compliance with the therapy.
28. At high risk of having a medical complication from the endoscopic procedure or Aspiration Therapy weight loss program for any reason, including poor general health or severe organ dysfunction, such as cirrhosis or renal dysfunction (GFR <60 mL/min/1.73 m2 at screening, calculated by using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2012-11-13 (Actual); Primary Completion 2015-06-24 (Actual); Study Completion 2019-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Thompson, MS, MD, Principal Investigator — Brigham and Women's Hospital
Locations (10):
- United States (10):
  - Dept VA San Diego Health Care System, San Diego, California
  - Howard University Center for Wellness and Weight Loss Surgery, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - University of Pennsylvania Center for Weight and Eating Disorders, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.

REFERENCES:
- See also: Aspire Bariatrics, Inc. Study Sponsor Website — http://www.aspirebariatrics.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject Screened Oct 30, 2012; First Subject Enrolled Nov 13, 2012; Last Subject Enrolled June 13, 2014
Period: Overall Study
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Started | 111 | 60
Completed | 82 | 31
Not Completed | 29 | 29
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 0 | 10
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 18 | 16
Not completed — Moved from area | 5 | 0
Not completed — medical - unrelated | 1 | 2
Not completed — nausea / discomfort | 3 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspiration Therapy | Lifestyle Therapy | Total
Number analyzed (Participants) | 111 | 60 | 171
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 111 | 60 | 171
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (10.0) | 46.8 (11.6) | 43.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 53 | 149
  Male | 15 | 7 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 99 | 49 | 148
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 17 | 50
  White | 74 | 42 | 116
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 111 | 60 | 171
Baseline Weight [Mean (Standard Deviation); unit: Kilograms] | 116.9 (21.2) | 112.8 (16.1) | 115.4 (19.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Excess Weight Loss (%EWL)
Description: The first effectiveness co-primary endpoint is the mean percent excess weight loss (%EWL) at 52-weeks. The hypothesis for the first primary effectiveness endpoint is that the difference in the mean percent excess weight loss (%EWL) at 52-weeks for the Aspiration Therapy (AT) group and Control group is at least 10%. Percent EWL is defined as absolute weight loss divided by baseline excess weight and multiplied by 100. Excess weight is determined from ideal body weights based on a BMI=25 kg/m2.
Time Frame: 52 weeks
Population: Modified Intent To Treat (mITT) population defined as all enrolled subjects
Measure: Mean (Standard Deviation); unit: Percent Excess Weight Loss
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Number analyzed (Participants) | 111 | 60
Percent Excess Weight Loss | 31.5 (26.7) | 9.8 (15.5)

2. Primary Outcome: % of Subjects Who Achieve >25% EWL
Description: The second co-primary effectiveness endpoint is that at least 50% of the AT group at 52-weeks achieve > 25% EWL.
Time Frame: 52 weeks
Population: Modified Intent To Treat (mITT) population of all enrolled subjects
Measure: Number (95% Confidence Interval); unit: Percent of Subjects
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Number analyzed (Participants) | 111 | 60
Percent of Subjects | 56.8 [49.0 to 64.5] | 22.0 [15.3 to 28.1]

3. Secondary Outcome: Mean Percent Total Body Weight Loss
Description: i) Mean percent absolute weight loss in AT compared to Control group
Time Frame: 52 weeks
Population: Modified Intent To Treat (mITT) population of all enrolled subjects
Measure: Mean (Standard Deviation); unit: Percent Total Weight Loss
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Number analyzed (Participants) | 111 | 60
Percent Total Weight Loss | 12.1 (9.6) | 3.6 (6.0)

4. Secondary Outcome: Percent of Subjects With ≥10% Total Body Weight Loss
Description: ii) proportion of subjects who achieve ≥10% absolute weight loss in AT compared to Control group
Time Frame: 52 weeks
Population: Modified Intent To Treat (mITT) population of all enrolled subjects
Measure: Number (95% Confidence Interval); unit: Percent of Subjects
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Number analyzed (Participants) | 111 | 60
Percent of Subjects | 58.6 [50.3 to 66.6] | 11.9 [5.7 to 21.1]

5. Secondary Outcome: Mean Percent Change in Serum Lipids
Description: iii) mean percent change serum lipids (triglyceride, HDL-cholesterol and LDL-cholesterol concentration) in the AT group compared to the control group
Time Frame: 52 weeks
Population: Subjects who completed 52 weeks
Measure: Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Number analyzed (Participants) | 82 | 31
Percent Change
  High Density Lipoprotein | 8.1 [4.2 to 12.0] | 1.7 [-3.8 to 7.2]
  Low Density Lipoprotein | -4.2 [-8.5 to 0.1] | -1.8 [-8.8 to 5.2]
  Triglycerides | -9.9 [-17.7 to -2.0] | 0.1 [-15.9 to 16.1]

6. Secondary Outcome: Mean Percent Change in Blood Pressure
Description: iv) mean percent change in systolic and diastolic blood pressures in the AT group compared to the control group
Time Frame: 52 weeks
Population: Subjects who completed 52 weeks
Measure: Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Number analyzed (Participants) | 82 | 31
Percent Change
  Systolic Pressure | -1.2 [-4.0 to 1.5] | -2.5 [-5.9 to 0.9]
  Diastolic Pressure | -2.6 [-5.2 to 0.1] | 0.5 [-4.1 to 5.2]

7. Secondary Outcome: Mean Change in Score for IWQOL Questionnaire
Description: v) "Impact of Weight on Quality of Life" (IWQOL) questionnaire total score
  Total score ranges from a minimum of 0 to a maximum of 100. Based on the algorithm developed by Crosby, et.al., patients' IWQOLLite total scores are considered to have shown meaningful improvement from baseline to one year if they increased between 7 and 12 points, depending upon baseline severity in comparison to the normative mean. Normative means for the IWQOL-Lite have been derived from a sample of 534 non-obese individuals who were not enrolled in any weight loss treatment program [238 women and 296 men with BMI's between 18.5 and 29.9]. The data presented is the mean change in total score. The AT group demonstrated a mean improvement (increase) in score of 16.3 points, the Control group a mean improvement (increase) of 11.7 points.
Time Frame: 52 weeks
Population: Subjects who completed the Questionnaire at 52 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Number analyzed (Participants) | 81 | 27
score on a scale | 16.3 [12.5 to 20.1] | 11.7 [5.5 to 17.9]

8. Secondary Outcome: Mean Change in Hemoglobin A1C
Description: vi) change in mean hemoglobin A1C (only subjects with T2 diabetes at baseline). Hemoglobin A1C is measured as DCCT%. The change in mean DCCT% from Baseline to Week 52 is reported for this secondary endpoint.
Time Frame: 52 weeks
Population: Subjects with Type 2 Diabetes
Measure: Mean (95% Confidence Interval); unit: DCCT% change
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Number analyzed (Participants) | 2 | 3
DCCT% change | -2.3 [-3.7 to -0.9] | -0.37 [-0.77 to -0.03]

9. Secondary Outcome: Procedural Success
Description: vii) percent procedural success (defined as successful endoscopic placement of the A-Tube) in all subjects undergoing endoscopy
Time Frame: 52 weeks
Population: All A-Tube placement attempts
Measure: Number; unit: Percent Procedural Success
Arm/Group | Aspiration Therapy
Number analyzed (Participants) | 112
Percent Procedural Success | 99

10. Secondary Outcome: Change in Medication for Hypertension
Description: Percent change in the number of medications taken by subjects for hypertension
Time Frame: 52 weeks
Population: Subjects being treated with medications for hypertension
Measure: Number; unit: Percent Change in Medications
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Number analyzed (Participants) | 29 | 20
Percent Change in Medications | -53.5 | -9.4

11. Secondary Outcome: Change in Medications for Dyslipidemia
Description: Percent change in the number of medications taken by subjects for dyslipidemia
Time Frame: 52 weeks
Population: Subjects being treated for high cholesterol
Measure: Number; unit: Percent Change in Medications
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Number analyzed (Participants) | 13 | 12
Percent Change in Medications | -23.1 | -7.7

12. Secondary Outcome: Change in Medications for Type 2 Diabetes
Description: Percent change in the number of medications taken by subjects for Type 2 Diabetes
Time Frame: 52 weeks
Population: Subjects being treated for Type 2 Diabetes
Measure: Number; unit: Percent Change in Medications
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Number analyzed (Participants) | 3 | 6
Percent Change in Medications | -33.0 | -14.3

13. Secondary Outcome: Change in Number of Subjects on Hypertension Medication
Description: Percent change in the number of subjects on Hypertension medication
Time Frame: 52 weeks
Population: Subjects being treated for hypertension
Measure: Number; unit: % Change in Subjects on Medication
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Number analyzed (Participants) | 29 | 20
% Change in Subjects on Medication | -62.1 | -10.0

14. Secondary Outcome: Change in Number of Subjects on Dyslipidemia Medications
Description: Percent change in the number of subjects on Dyslipidemia medications
Time Frame: 52 weeks
Population: Subjects being treated for high cholesterol
Measure: Number; unit: % Change in Subjects on Medication
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Number analyzed (Participants) | 13 | 12
% Change in Subjects on Medication | -23.1 | -8.3

15. Secondary Outcome: Change in Number of Subjects on Diabetes Medication
Description: Percent change in the number of subjects on Diabetes medication
Time Frame: 52 weeks
Population: Subjects being treated for Type II Diabetes
Measure: Number; unit: % Change in Subjects on Medication
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Number analyzed (Participants) | 3 | 6
% Change in Subjects on Medication | -33.3 | -16.7

16. Other Pre Specified Outcome: Safety Outcomes
Description: The incidence of procedure-related, device-related, and therapy-related serious adverse events. Also, the development of adverse eating behaviors will be assessed.
Time Frame: 52 weeks
Population: Modified Intent To Treat (mITT) population of all enrolled subjects
Measure: Number; unit: Percent of Subjects
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Number analyzed (Participants) | 111 | 60
Percent of Subjects
  Serious Adverse Event | 3.6 | 0
  Diagnosed Eating Disorder | 0 | 1.7

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Aspiration Therapy | Lifestyle Therapy
Serious Adverse Events (participants affected / at risk) | 4/111 | 0/60
Other Adverse Events (participants affected / at risk) | 93/111 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspiration Therapy (N=111) | Lifestyle Therapy (N=60)
Peritonitis (Surgical and medical procedures) | 1 (1) | 0 (0) — Peritonitis (mild pneumo-peritoneum without abscess) post endoscopic A-Tube placement
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 0 (0) — Abdominal pain post endoscopic A-Tube placement procedure
Prepyloric Ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) — Non-bleeding pre-pyloric ulceration
A-Tube Replacement (Surgical and medical procedures) | 1 (1) | 0 (0) — A-Tube replaced, Site documented as SAE because endoscopy was performed to replace the tube.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspiration Therapy (N=111) | Lifestyle Therapy (N=60)
Granulation Tissue (Skin and subcutaneous tissue disorders) | 45 (45) | 0 (0) — Granulation tissue at the stoma site is a normal healing process but can cause discomfort if not treated.
Abdominal Pain (post procedure) (Gastrointestinal disorders) | 42 (42) | 0 (0) — Abdominal pain occurring within 4 weeks of the A-Tube endoscopic placement
Peristomal Discharge (Skin and subcutaneous tissue disorders) | 34 (34) | 0 (0) — Peristomal bleeding, discharge, inflammation, irritation
Nausea / Vomiting (Gastrointestinal disorders) | 21 (21) | 0 (0) — Nausea and vomiting generally the result of sedation and post procedure pain medication
Abdominal Discomfort (Gastrointestinal disorders) | 21 (21) | 0 (0) — Intermittent abdominal discomfort
Peristomal Infection (Infections and infestations) | 16 (16) | 0 (0) — Peristomal bacterial infection / possible infection
Abdominal Pain (after 4 weeks) (Gastrointestinal disorders) | 9 (9) | 0 (0) — Abdominal pain onset more than 4 weeks after A-Tube placement
Change in Bowel Habits (Gastrointestinal disorders) | 5 (5) | 0 (0) — Dyspepsia, Constipation, Diarrhea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No